CLINICAL TRIAL: NCT03920527
Title: A Randomized Controlled Trial to Compare the Clinical Outcomes of Six Months Versus 12 Months of Oral Itraconazole Therapy for Management of Treatment naïve Subjects With Chronic Pulmonary Aspergillosis
Brief Title: Six Months Versus 12 Months of Oral Itraconazole Therapy for Management of Treatment naïve Subjects With CPA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Inderpaul singh, Assistant Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NK/4947/Res/986
Record Dates: First submitted 2019-04-09; First posted 2019-04-19 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Chronic Pulmonary Aspergillosis
Keywords: CPA; Aspergillosis; CCPA; CFPA
MeSH Terms: conditions — Aspergillosis | interventions — Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Six months (Active Comparator): Six months of itraconazole
  Interventions: Drug: Itraconazole 400 mg
- 12 months (Experimental): 12-months of itraconazole
  Interventions: Drug: Itraconazole 400 mg

INTERVENTIONS:
Drug: Itraconazole 400 mg — Duration of itraconazole
  Other Names: sporanox

SUMMARY:
The treatment options majorly consist of medical management with at least 6-month long treatment with antifungal drugs - most significantly the azole groups. Itraconazole is the preferred azole for the treatment of CPA. The duration of treatment with oral itraconazole remains uncertain. In a previous study the use of oral itraconazole for 6-months a favorable overall response was seen in 76% of the subjects. Moreover, about 30%-50% of the subjects have disease relapse that requires prolonged therapy. It is likely that a longer duration of itraconazole would have a higher response rate and thus, lower risk of relapse after discontinuation of therapy. In this randomized controlled trial, we compare the clinical outcomes of six months versus twelve months of itraconazole therapy in treatment naïve subjects with chronic pulmonary aspergillosis

DETAILED DESCRIPTION:
Aspergillus is a saprophytic fungus which is present normally in our surroundings and causes a large number of pulmonary diseases spreading through inhalational route. The spectrum of disease caused by aspergillus spp. is wide with the manifestations of the disease being governed primarily by the status of the underlying host immunity, which then determines the nature of the host-aspergillus interaction. Patients with an intact immunity have a more stable and indolent form of disease like aspergilloma whereas with a worsening immune status, the risk of invasive disease increases. Chronic pulmonary aspergillosis (CPA) and allergic bronchopulmonary aspergillosis (ABPA) are two of the commonest pulmonary manifestations seen in non-immunocompromised patients whereas invasive pulmonary aspergillosis being more common in the immunocompromised patients.

Estimates suggest that CPA affects around 3 million people across the globe, which may still be an under estimated number as the disease co exists with other pulmonary co-morbidities which make accurate diagnosis a pitfall. In India the annual incidence of CPA was estimated in 2011 and varied between 27,000-0.17 million cases, with different estimates. Based on the mortality rate for CPA which was estimated to be 15% annually, the 5-year prevalence of CPA was placed at 290,147 cases with 5-year prevalence rate being 24 per 100,000 in the same year. The disease confers significant morbidity and mortality, making it a significant burden for the society as well as the healthcare. Apart from the respiratory symptoms, CPA causes significant constitutional symptoms as well which adds to the misery of the patient. The diagnosis of CPA is based on presence of chronic symptoms, consistent radiology and demonstration of Aspergillus by direct (culture) or indirect (serological) methods. Even though CPA is more of a disease spectrum but overall it is characterized by slowly progressive lung cavitation which may or may not show presence of mycetoma /fungal ball in patients with pre-existing structural lung diseases, even though other patterns have also been identified.

The treatment options majorly consist of medical management with at least 6-month long treatment with antifungal drugs - most significantly the azole groups. Itraconazole is the preferred azole for the treatment of CPA. The duration of treatment with oral itraconazole remains uncertain. In a previous study the use of oral itraconazole for 6-months a favorable overall response was seen in 76% of the subjects. Moreover, about 30%-50% of the subjects have disease relapse that requires prolonged therapy. It is likely that a longer duration of itraconazole would have a higher response rate and thus, lower risk of relapse after discontinuation of therapy. In this randomized controlled trial, we compare the clinical outcomes of six months versus twelve months of itraconazole therapy in treatment naïve subjects with chronic pulmonary aspergillosis.

ELIGIBILITY:
Inclusion Criteria: includes presence of all the following:

* one or more clinical symptoms (persistent cough, recurrent hemoptysis, weight loss, malaise, fever and dyspnea) for ≥3 months
* slowly progressive or persistent radiological findings (one or more cavities and surrounding fibrosis, infiltrates, consolidation, with or without fungal ball or progressive pleural thickening) on computed tomography (CT) of the thorax
* immunological (A.fumigatus-specific IgG >27 mgA/L or positive Aspergillus precipitins) or microbiological evidence of Aspergillus infection (growth of Aspergillus in respiratory secretions or serum galactomannan index >0.5 or BALF galactomannan index >1) and,
* exclusion of other pulmonary disorders with similar presentation.

Exclusion Criteria:

* failure to provide informed consent
* patients on immunosuppressive drugs, intake of prednisolone (or equivalent) >10 mg for at least 3 weeks or a diagnosis of human immunodeficiency virus syndrome
* intake antifungal azoles for >3 weeks in the preceding six months
* subjects with active pulmonary infection due to mycobacterium tuberculosis or mycobacteria other than tuberculosis (MOTT)
* subjects with others forms of pulmonary aspergillosis (allergic bronchopulmonary aspergillosis, chronic necrotizing aspergillosis and angio-invasive aspergillosis)
* pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-08-15 (Actual)

PRIMARY OUTCOMES:
Relapse rate | 2 year after randomization
  number of relapses at 2 year after randomization

SECONDARY OUTCOMES:
Response | at 6 to 12 months
  Proportion of subjects with an overall favourable response at the end of oral itraconazole therapy
Adverse events | 1 year
  adverse events due to itraconazole

CONTACTS AND LOCATIONS:
Locations (1):
- Inderpaul Singh, Chandigarh, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sehgal IS, Dhooria S, Muthu V, Prasad KT, Aggarwal AN, Chakrabarti A, Choudhary H, Garg M, Agarwal R. Efficacy of 12-months oral itraconazole versus 6-months oral itraconazole to prevent relapses of chronic pulmonary aspergillosis: an open-label, randomised controlled trial in India. Lancet Infect Dis. 2022 Jul;22(7):1052-1061. doi: 10.1016/S1473-3099(22)00057-3. Epub 2022 Apr 13. PMID 35429465